CLINICAL TRIAL: NCT00000199
Title: Piracetam for Treatment of Cocaine Addiction, Phase II
Brief Title: Piracetam for Treatment of Cocaine Addiction, Phase II - 4
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-00238-4; K20DA000238 (NIH); K02-00238-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Piracetam

INTERVENTIONS:
Drug: Piracetam

SUMMARY:
The purpose of this study is to follow patients in Phase I of an inpatient study in an eight week open label assessment of piracetam in an outpatient treatment program.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Drug use
Adverse effects
Clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Kampman, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States